CLINICAL TRIAL: NCT04568889
Title: Minnesota COVID-19 Testing Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Abdul Latif Jameel Poverty Action Lab (Other); Government of Minnesota Office of Management and Budget (Unknown)
Responsible Party: Principal Investigator, Marcella Alsan, Professor, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB20-1444
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Covid19; Infectious Disease
Keywords: COVID-19; Minnesota; Unit nonresponse; Item nonresponse
MeSH Terms: conditions — COVID-19; Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Government/High Incentive/Cost-Benefit Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $20 incentive. Then the participant is assigned to be a message that emphasizes the public health benefits of answering the survey questions (i.e. cost-benefit frame).
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: Cost-Benefit Frame
- Government/High Incentive/Duty Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $20 incentive. Then the participant is assigned to be a message that emphasizes an individual's responsibility to their community (i.e. duty frame).
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: Duty Frame
- Government/High Incentive/Racial/Ethnic Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $20 incentive. Then the participant is assigned to be a message that emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups.
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: Racial/Ethnic Frame
- Government/High Incentive/No Message Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $20 incentive. Then the participant is assigned to the arm that provides no messaging.
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: No Messaging
- Researchers/High Incentive/Cost-Benefit Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $20 incentive. Then the participant is assigned to be a message that emphasizes the public health benefits of answering the survey questions (i.e. cost-benefit frame).
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: Cost-Benefit Frame
- Researchers/High Incentive/Duty Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $20 incentive. Then the participant is assigned to be a message that emphasizes an individual's responsibility to their community (i.e. duty frame).
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: Duty Frame
- Researchers/High Incentive/Racial/Ethnic Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $20 incentive. Then the participant is assigned to be a message that emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups.
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: Racial/Ethnic Frame
- Researchers/High Incentive/No Message Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $20 incentive. Then the participant is assigned to the arm that provides no messaging.
  Interventions: Behavioral: A $20 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: No Messaging
- Government/Low Incentive/Cost-Benefit Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $10 incentive. Then the participant is assigned to be a message that emphasizes the public health benefits of answering the survey questions (i.e. cost-benefit frame).
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: Cost-Benefit Frame
- Government/Low Incentive/Duty Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $10 incentive. Then the participant is assigned to be a message that emphasizes an individual's responsibility to their community (i.e. duty frame).
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: Duty Frame
- Government/Low Incentive/Racial/Ethnic Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $10 incentive. Then the participant is assigned to be a message that emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups.
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: Racial/Ethnic Frame
- Government/Low Incentive/No Message Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing government involvement and a $10 incentive. Then the participant is assigned to the arm that provides no messaging.
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Government Involvement; Behavioral: No Messaging
- Researchers/Low Incentive/Cost-Benefit Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $10 incentive. Then the participant is assigned to be a message that emphasizes the public health benefits of answering the survey questions (i.e. cost-benefit frame).
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: Cost-Benefit Frame
- Researchers/Low Incentive/Duty Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $10 incentive. Then the participant is assigned to be a message that emphasizes an individual's responsibility to their community (i.e. duty frame).
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: Duty Frame
- Researchers/Low Incentive/Racial/Ethnic Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $10 incentive. Then the participant is assigned to be a message that emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups.
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: Racial/Ethnic Frame
- Researchers/Low Incentive/No Message Frame (Experimental): The participant is assigned to receive a flyer that includes a message emphasizing the involvement of academic researchers and a $10 incentive. Then the participant is assigned to the arm that provides no messaging.
  Interventions: Behavioral: A $10 Survey Incentive; Behavioral: Emphasis of Academic Researchers Involvement; Behavioral: No Messaging

INTERVENTIONS:
Behavioral: A $10 Survey Incentive — Individuals see a 10 dollar incentive on the flyers advertising the baseline survey.
  Arms: Government/Low Incentive/Cost-Benefit Frame; Government/Low Incentive/Duty Frame; Government/Low Incentive/No Message Frame; Government/Low Incentive/Racial/Ethnic Frame; Researchers/Low Incentive/Cost-Benefit Frame; Researchers/Low Incentive/Duty Frame; Researchers/Low Incentive/No Message Frame; Researchers/Low Incentive/Racial/Ethnic Frame
Behavioral: A $20 Survey Incentive — Individuals see a 10 dollar incentive on the flyers advertising the baseline survey.
  Arms: Government/High Incentive/Cost-Benefit Frame; Government/High Incentive/Duty Frame; Government/High Incentive/No Message Frame; Government/High Incentive/Racial/Ethnic Frame; Researchers/High Incentive/Cost-Benefit Frame; Researchers/High Incentive/Duty Frame; Researchers/High Incentive/No Message Frame; Researchers/High Incentive/Racial/Ethnic Frame
Behavioral: Emphasis of Government Involvement — Individuals see a message emphasizing the involvement of the government in the study,
  Arms: Government/High Incentive/Cost-Benefit Frame; Government/High Incentive/Duty Frame; Government/High Incentive/No Message Frame; Government/High Incentive/Racial/Ethnic Frame; Government/Low Incentive/Cost-Benefit Frame; Government/Low Incentive/Duty Frame; Government/Low Incentive/No Message Frame; Government/Low Incentive/Racial/Ethnic Frame
Behavioral: Emphasis of Academic Researchers Involvement — Individuals see a message emphasizing the involvement of academic researchers in the study,
  Arms: Researchers/High Incentive/Cost-Benefit Frame; Researchers/High Incentive/Duty Frame; Researchers/High Incentive/No Message Frame; Researchers/High Incentive/Racial/Ethnic Frame; Researchers/Low Incentive/Cost-Benefit Frame; Researchers/Low Incentive/Duty Frame; Researchers/Low Incentive/No Message Frame; Researchers/Low Incentive/Racial/Ethnic Frame
Behavioral: Cost-Benefit Frame — Individuals will see messaging that emphasizes the public health benefits of answering the survey questions in the baseline survey (cost-benefit frame).
  Arms: Government/High Incentive/Cost-Benefit Frame; Government/Low Incentive/Cost-Benefit Frame; Researchers/High Incentive/Cost-Benefit Frame; Researchers/Low Incentive/Cost-Benefit Frame
Behavioral: Duty Frame — Individuals will see messaging that emphasizes an individual's responsibility to their community in the baseline survey (duty frame),
  Arms: Government/High Incentive/Duty Frame; Government/Low Incentive/Duty Frame; Researchers/High Incentive/Duty Frame; Researchers/Low Incentive/Duty Frame
Behavioral: Racial/Ethnic Frame — Individuals will see messaging that emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups in the baseline survey.
  Arms: Government/High Incentive/Racial/Ethnic Frame; Government/Low Incentive/Racial/Ethnic Frame; Researchers/High Incentive/Racial/Ethnic Frame; Researchers/Low Incentive/Racial/Ethnic Frame
Behavioral: No Messaging — Individuals will see no messaging in the baseline survey.
  Arms: Government/High Incentive/No Message Frame; Government/Low Incentive/No Message Frame; Researchers/High Incentive/No Message Frame; Researchers/Low Incentive/No Message Frame

SUMMARY:
The goal of this project is to help the state of Minnesota understand why individuals are not getting tested and potentially identify trusted individuals or organizations that could be used in follow-up work to send messages. Investigators focus on the first two issues of unit and item nonresponse, which is not random across the population and thus could lead to nonresponse bias. To do so, investigators are deploying flyers through 10 Twin City area food shelves and potentially through public housing units with information on how to answer an online questionnaire.

DETAILED DESCRIPTION:
In the United States, recent statistics show that African American and Latinx communities bear a disproportionate burden from COVID-19. Reaching vulnerable and underserved populations is therefore crucial to combating the disease. However, most public messaging campaigns are not targeted toward underserved communities and don't address fears of social stigma, mistrust in the healthcare system, or concerns about immigration status.

The goal of this project is to help the state of Minnesota understand why individuals are not getting tested and potentially identify trusted individuals or organizations that could be used in follow-up work to send messages. To do so, investigators are deploying flyers through 10 Twin City area food shelves and potentially through public housing units with information on how to answer an online questionnaire.

This provides us with an opportunity to study who answers surveys and why - and what questions are particularly sensitive. This is of general interest to academicians and policymakers alike.

The quality of household surveys is in decline, for three main reasons. First, households have become increasingly less likely to answer surveys at all (unit nonresponse). Second, those that respond are less likely to answer certain questions (item nonresponse). Third, when households do provide answers, they are less likely to be accurate (measurement error). This is important since household surveys help to estimate the employment rate, healthcare needs and of course the census determines resources/representation.

Investigators focus on the first two issues of unit and item nonresponse, which is not random across the population and thus could lead to nonresponse bias. Census tracts with predominantly Hispanic or Black residents had significantly lower response rates to the American Community Survey as compared to the response rates in predominantly white tracts. Similarly, response rates to the Health Information National Trends Survey (HINTS) were lower in areas with higher levels of Hispanic and minority residents.

Investigators hypothesize that financial incentives may encourage unit response; conversely, a close association with the government may discourage response. To test these hypotheses, investigators plan to cross-randomize the incentive amount offered and the emphasis placed on government involvement in the study on flyers advertising the baseline survey. Individuals will see either a) a 10 dollar incentive, or b) a 20 dollar incentive; and either a) messaging that emphasizes government involvement in the study, or b) messaging that emphasizes the involvement of academic researchers. Flyers will be randomized at the foodshelf-day level.

To test what affects item non-response on potentially sensitive questions, such as questions which ask for health information, investigators hypothesize that ethical framing may encourage individuals to answer questions. This takes two forms --- the deontological (or duty based) frame, and the consequential (or cost-benefit) frame. Moreover, knowing others feel the same way (regarding the obligation or benefits of providing health information) may amplify motivation. Finally, there is the possibility that emphasizing the importance of ethnic and racial disadvantage associated with COVID-19 outcomes may be important for improving item non-response on sensitive questions.

Upon completion of the demographic module of the survey but prior to starting several potentially sensitive survey modules, individuals will see a message that either a) emphasizes the public health benefits of answering the survey questions (cost-benefit frame); b) emphasizes an individual's responsibility to their community (duty frame); c) emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups; or d) provides no messaging. Messaging content will be randomized at the individual level.

ELIGIBILITY:
Inclusion Criteria:

* All participants who are aged 18 or above and speak English or Spanish

Exclusion Criteria:

* Children, those who do not identify as above or adults who identify as above but do not agree to participate in survey during the consent stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Effect of monetary incentives in increasing unit response 1 | This outcome will be assessed when the individual agrees to participate in the Baseline survey, which takes approximately 20 minutes.
  Number of participants who received a flyer that mentions a $20 incentive and completed the survey
Effect of monetary incentives in increasing unit response 2 | This outcome will be assessed when the individual agrees to participate in the Baseline survey, which takes approximately 20 minutes.
  Number of participants who received a flyer that mentions a $10 incentive and completed the survey.
Effect of a government frame in reducing unit response 1 | This outcome will be assessed when the individual agrees to participate in the Baseline survey, which takes approximately 20 minutes.
  Number of participants who received a flyer that mentions a government frame and completed the survey
Effect of a government frame in reducing unit response 2 | This outcome will be assessed when the individual agrees to participate in the Baseline survey, which takes approximately 20 minutes.
  Number of participants who received a flyer that mentions a research frame and completed the survey.
Interactions between monetary incentives and a government frame 1 | This outcome will be assessed when the individual agrees to participate in the Baseline survey, which takes approximately 20 minutes.
  Number of participants who received a flyer that mentions a government frame and $20 incentive and completed the survey
Interactions between monetary incentives and a government frame 2 | This outcome will be assessed when the individual agrees to participate in the Baseline survey, which takes approximately 20 minutes.
  Number of participants who received a flyer that mentions a government frame and $10 incentive and completed the survey
Interactions between monetary incentives and a government frame 3 | This outcome will be assessed during the 20-minute Baseline Survey.
  Number of participants who received a flyer that mentions a researcher frame and $20 incentive and completed the survey
Interactions between monetary incentives and a government frame 4 | This outcome will be assessed during the 20-minute Baseline Survey.
  Number of participants who received a flyer that mentions a researcher frame and $10 incentive and completed the survey
Demographic characteristics of participants assigned into each treatment arm | This outcome will be assessed during the 20-minute Baseline Survey.
  Demographic characteristics (e.g. sex, education level, income level, race/ethnicity) of participants who are assigned to each treatment arm and completed the survey.
Effect of various messaging frames in increasing item non-response | This outcome will be assessed during the 20-minute Baseline Survey.
  Number of survey participants who are randomly assigned to receive each messaging frame that: a) emphasizes the public health benefits of answering the survey questions (cost-benefit frame); b) emphasizes an individual's responsibility to their community (duty frame); c) emphasizes the disproportionate impact of COVID-19 on certain ethnic and racial groups; or d) provides no messaging.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella Alsan, MD, MPH, PhD, Principal Investigator — Harvard Kennedy School
Locations (10):
- United States (10):
  - Volunteers Enlisted to Assist People, Bloomington, Minnesota
  - Southern Anoka Community Assistance, Columbia Heights, Minnesota
  - People Reaching Out to People Food Shelf, Eden Prairie, Minnesota
  - Fridley Covenant Church, Fridley, Minnesota
  - Calvary Lutheran Church Food Shelf, Minneapolis, Minnesota
  - NorthPoint Health and Wellness, Minneapolis, Minnesota
  - Community Emergency Assistance Programs, Minneapolis, Minnesota
  - Intercongregation Communities Association, Minnetonka, Minnesota
  - Valley Outreach, Stillwater, Minnesota
  - White Bear Area Foodshelf, White Bear Lake, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffin, DH. Measuring survey nonresponse by race and ethnicity. In Proceedings of the Annual Meetings of the American Statistical Association. 2002; 11-15.
- [Background] Maitland A, Lin A, Cantor D, Jones M, Moser RP, Hesse BW, Davis T, Blake KD. A Nonresponse Bias Analysis of the Health Information National Trends Survey (HINTS). J Health Commun. 2017 Jul;22(7):545-553. doi: 10.1080/10810730.2017.1324539. Epub 2017 May 30. PMID 28557627
- [Result] Meyer, Bruce D., Wallace KC Mok, and James X. Sullivan. Household surveys in crisis. Journal of Economic Perspectives. 2015; 29(4): 199-226.

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT04568889/SAP_000.pdf